CLINICAL TRIAL: NCT01501318
Title: Brief Education to Reduce Health Care Consumers' Risky Substance Use Behaviors: How Brief is Brief?
Brief Title: Impact of Personalized Feedback Alone on Substance Use Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of Missouri, St. Louis (Other); Institute of Mental Health, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1200450
Record Dates: First submitted 2011-12-23; First posted 2011-12-29 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Substance Abuse
Keywords: SBIRT; brief intervention; alcohol; drug abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized feedback plus education (Active Comparator): Participants receive the personalized feedback report plus education. This is the currently implemented service approach.Treatment as usual with participants receiving a personalized feedback report about the risks associated with their current substance use behaviors and a brief (5-15 minute) motivational interviewing based education session provided by a trained health coach.
  Interventions: Behavioral: Personalized feedback report plus education
- Personalized feedback report alone (Experimental): Provision of the personalized feedback report alone.
  Interventions: Behavioral: Personalized feedback report

INTERVENTIONS:
Behavioral: Personalized feedback report — Participants receive the personalized feedback report but no additional education.
  Arms: Personalized feedback report alone
Behavioral: Personalized feedback report plus education — Participants receive the personalized feedback report plus education. This is the currently implemented service approach.
  Arms: Personalized feedback plus education

SUMMARY:
The investigators seek to develop a more efficient and effective approach to providing brief behavioral health interventions for risky substance use behaviors by comparing a brief coach directed intervention to a tailored report only group.

DETAILED DESCRIPTION:
Screening and brief intervention (SBIRT) generally involves universal screening for risky substance use behaviors in medical settings and the immediate provision of a 3-15 minute intervention to those found to be at risk. In this pilot study, the investigators seek to develop a more efficient and effective approach to providing brief behavioral health interventions in the field by comparing a brief coach directed intervention to a tailored report only group. The goal is to create a cost-effective and sustainable system that provides consumers with tailored information that will help them both initiate and sustain the lifestyle changes necessary for improving their overall health.

Hypothesis 1: In a medical setting, personalized feedback alone will be associated with a reduction in risky substance use behaviors.

Hypothesis 2: In a medical setting, personalized feedback alone will have the same impact on behavior as that information plus a brief coach education session on risky substance use behaviors..

ELIGIBILITY:
Inclusion Criteria:

* Low level risky substance use

Exclusion Criteria:

* high substance use risk levels
* potential alcohol or drug addiction or dependence

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Substance use behaviors and consequences | 1 month follow-up
  Interview questionnaire includes items concerning substance use behaviors (e.g., the number of drinks in the last 7 days) and consequences {e.g., ''During the past month, how often have you failed to do what was normally expected of you because of your use of alcohol?'

SECONDARY OUTCOMES:
Substance use behavioral intentions | 1 month follow-up
  Interview questionnaire that asks participants about their memory of the materials provided in the intervention, their motivation toward change, and their self-reported change efforts.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew G Hile, PhD, Principal Investigator — Missouri Institute of Mental Health
Locations (1):
- University of Missouri Hospital ER, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No